CLINICAL TRIAL: NCT05893667
Title: Evaluation of Pretreatment Inflammatory Markers in Predicting Response to nCRT and Prognosis in LARC Patients
Brief Title: Evaluation of Inflammatory Markers in LARC Patients
Status: Completed | Type: Observational
Sponsor: Hospital Pedro Hispano (Other)
Responsible Party: Principal Investigator, Marina Morais, Principal Investigator, Hospital Pedro Hispano
Other Study IDs: HPedroHispano
Record Dates: First submitted 2023-05-17; First posted 2023-06-08 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Locally Advanced Rectal Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High levels of inflammatory scores
  Interventions: Diagnostic Test: Inflammatory markers
- Low levels of inflammatory scores
  Interventions: Diagnostic Test: Inflammatory markers

INTERVENTIONS:
Diagnostic Test: Inflammatory markers — analysis of inflammatory scores

SUMMARY:
Introduction: In locally advanced rectal cancers (LARC), TNM staging is far from optimal. We aimed to investigate the value of previously described circulating biomarkers as predictors of prognosis.

Methods: Retrospective analysis of 245 LARC patients diagnosed between January 2010 and December 2022, who underwent neoadjuvant chemoradiotherapy and surgery at two centers. A Cox regression and Kaplan-Meier analysis were performed.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed pathologically with rectal adenocarcinomas, located within 12cm from the anal verge (measured by MRI), clinically staged T3-4 and/or N+ and treated with neoadjuvant chemoradiotherapy (nCRT) followed by radical surgery

Exclusion Criteria:

* evidence of distant metastasis at diagnosis, emergent or palliative surgery, local excision or "watch and wait" approach and evidence of inflammatory or hematological disorders

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: as in inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 245 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Overall survival Disease-free survival | 5 years

SECONDARY OUTCOMES:
Pathological response through Ryan Tumor Regression Grade | at study completion, average of 5 years
  TRG 1-5; 1- no viable cancer cells; 5- no fibrosis, with extensive residual disease

IPD SHARING:
Plan to Share IPD: Undecided